CLINICAL TRIAL: NCT01051245
Title: Effectiveness of a High-risk Diabetic Patients Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Gaston Perman, Head of Medical Programs, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1494
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2 [C18.452.394.750.149]; Case Management [N04.590.233.624.250]; Disease Management [N04.590.607]; Diabetes Complications [C19.246.099]
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case management (Active Comparator): Patients followed-up by case manager. Interventions based on the Chronic Care Model. Interventions are self management education, motivational interviewing, individualized counseling on non-pharmacological treatment to modify and sustain healthy lifestyle behaviours, and follow-up. Close contact with primary care physician and/or specialist by case manager, if clinical targets out of recommended standards. Pharmacological treatment not suggested, managed by personal criteria of health care professionals. Focus on targets.
  Interventions: Behavioral: Case manager counseling
- Usual care group (Placebo Comparator): Usual care provided by primary care physician and/or specialist. Free access to diabetes educational workshops. Regular delivery of educational brochures (not personally targeted).
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Case manager counseling — Patients followed-up by case manager. Interventions based on the Chronic Care Model. Interventions are self management education, motivational interviewing, individualized counseling on non-pharmacological treatment to modify and sustain healthy lifestyle behaviours, and follow-up. Close contact with primary care physician and/or specialist by case manager, if clinical targets out of recommended standards. Pharmacological treatment not suggested, managed by personal criteria of health care professionals. Focus on targets.
  Arms: Case management
Other: Usual care — Usual care provided by primary care physician and/or specialist according to patients' needs and professional criteria. Includes free access to educational diabetes workshops and educational brochures.
  Arms: Usual care group

SUMMARY:
The purpose of this study is to determine whether case management for type 2 diabetic patients with target-organ damage improves quality of care compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus
* Age between 18 and 80 years old
* Target organ damage (either macrovascular or microvascular)
* Patient's acceptance to participate

Exclusion Criteria:

* Moderate to severe dementia
* Life expectancy lower than one year
* Justified negative from primary care physician to intervene the patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2010-03; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Combined outcome assessing adequate control of hypertension, LDL-cholesterol and glycated hemoglobin | Two years

SECONDARY OUTCOMES:
Quality of care process measures | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Gastón Perman, MD, MSc, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina